CLINICAL TRIAL: NCT07205302
Title: Safety and Efficacy of the Flow Diverter in the Treatment of Intracranial Non-saccular Aneurysm
Acronym: SAEFD
Status: Not yet recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RJSW202504
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Intracranial Non-saccular Aneurysms
Keywords: intracranial non-saccular aneurysms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year

GROUPS / COHORTS (1):
- FD: treatment of intracranial non-saccular aneurysms with flow diverter
  Interventions: Device: flow diverter

INTERVENTIONS:
Device: flow diverter — the treatment of intracranial non-saccular aneurysms with flow diverter

SUMMARY:
Using data obtained from the treatment of intracranial non-saccular aneurysms with flow diverter, evaluate the effecy and safety of blood flow diverter for the endovascular treatment of intracranial non-saccular aneurysms.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 80 years, any gender
2. Diagnosed as a non-saccular aneurysm in the patient's intracranial region
3. Subject or guardian is able to understand the purpose of study, shows sufficient compliance with the study protocol and provides a signed informed consent form

Exclusion Criteria:

1. Aneurysm rupture within 30 days before enrollment;
2. Diagnosis of multiple aneurysms and requiring reoperation within 12 months
3. Conditions that are not appropriate for stent delivery and deployment judged by investigators (severe stenosis of parent artery, severe tortuosity of parent artery, stent failing to reach the lesion, stent in the target lesion of parent artery, etc.);
4. Heart, lung, liver and renal failure or other severe diseases (intracranial tumor, systemic infection, disseminated intravascular coagulation, myocardial infarction within 12 months before enrollment, history of severe psychosis, severe stenosis or occlusion of cerebral feeding artery, etc.);
5. Major surgery within 30 days before enrollment，or planned to undergo surgery within 360 days after enrollment;
6. Known allergies or contraindications to anesthetics, anticoagulants, and antiplatelet drugs;
7. Known allergy to nickel-titanium alloy metal materials;
8. Life expectancy <12 months;
9. Pregnant or breastfeeding women;
10. Subject has participated in other clinical trials within 1 month before signing informed consent;
11. Other conditions judged by the investigators as unsuitable for enrollment.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with intracranial Non-saccular aneurysm
Sampling Method: Non-Probability Sample
Enrollment: 168 (Estimated)
Dates: Start 2025-10-08 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete occlusion rate of aneurysm 12 months after surgery | 12 months after surgery
  Complete occlusion is defined as no significant blood flow ,and achieves Raymond-Roy class I , which is diagnosed by cerebrovascular DSA at 6 months post-procedure.

IPD SHARING:
Plan to Share IPD: Undecided